CLINICAL TRIAL: NCT05780242
Title: Psychiatry and Anthropology Research Protocol : Recrudescence of Eating Conduct Disorders and Covid-19: a Qualitative Study for a Psychiatric and Anthropological Cross-view
Brief Title: Recrudescence of Eating Conduct Disorders and Covid-19
Acronym: TCA-Covid19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 22-HPNCL-06
Record Dates: First submitted 2023-03-20; First posted 2023-03-22 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-03

CONDITIONS: Psychiatric Disorder; Eating Disorders in Adolescence; COVID-19
MeSH Terms: conditions — Mental Disorders; COVID-19 | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TCA: interviews based on a questionnaire established beforehand evoking the history of eating disorders and the experience of the participant
  Interventions: Behavioral: Self-questionnaire Eating Attitudes; Behavioral: Situational Anxiety and Trait Anxiety; Behavioral: Beck Depression Inventory (BDI) scale; Behavioral: • Post-traumatic Check List Scale

INTERVENTIONS:
Behavioral: Self-questionnaire Eating Attitudes — self-diagnostic and quantitative questionnaire of 40 questions evaluating the behavior, severity and evolution of anorexia nervosa
Behavioral: Situational Anxiety and Trait Anxiety — assess anxiety as a "personality trait" (feelings of apprehension, tension, nervousness and worry that the subject usually feels), and anxiety as a ' "emotional state" linked to a particular situation
Behavioral: Beck Depression Inventory (BDI) scale — a diagnostic self-questionnaire allowing a quantitative estimation of the intensity of depressive symptoms in adults and adolescents
Behavioral: • Post-traumatic Check List Scale — questionnaire includes 20 items, each question is to be rated between 1 and 5 depending on the intensity and frequency of symptoms during the previous month.

SUMMARY:
This qualitative study, combining psychiatric and anthropological perspectives, focused on the development and/or worsening of patients' eating disorders since Covid-19, as well as the experiences and perceptions of those around them - such as their family, teachers or staff. School and nursing staff. This multi-site approach will provide a multidimensional perspective on the experience of individuals and those around them, as well as a triangulation of data. The hypotheses to explain the increase in Eating Disorders (EDs) will be addressed through semi-structured interviews offered to study participants.

DETAILED DESCRIPTION:
This study will be offered to all patients treated within the SUPEA of HPNCL for TCA. The active queue of patients is collected using the HPNCL medical software. Patients and their parents will be contacted by telephone to inform them and suggest that they participate in this study.

The schools will be chosen from those attended by the patients on this list. They will also be contacted by telephone to inform them and suggest that they participate in this study.

Interviews in the presence of two members of the research team (child psychiatrists, psychologists, anthropologists, etc.) will be offered to all patients. These interviews will be face-to-face when possible, but can also be done remotely, by teleconsultation, depending on the preferences of the participants.

These interviews will be based on a questionnaire established beforehand evoking the history of eating disorders and the experience of the participant in the study and his entourage of the Covid-19 health crisis.

All information exchanged during these interviews will be made anonymous (data collected and processed as well as the results presented). They will be used exclusively in the context of the study and not communicated to the medical team involved in the patient's care.

The proposed interviews will be carried out separately with:

* The patient presenting or having presented a TCA
* The parents
* One or more health professionals taking care of the patient
* The school attended by the patient who will be questioned about the TCA and Covid-19 problem in general or not about the patient in particular.

Questionnaires will also be carried out with patients in order to complete the assessment of their clinical condition at a distance from the psychological crisis:

ELIGIBILITY:
Inclusion Criteria:

Any patient having consulted in the child psychiatric emergency room of the HPNCL between November 1, 2021 and November 30, 2021 for suicidal thoughts.

Age between 13 years and 17 years and 11 months. Good understanding of written and oral French. Collection of the informed consent of the patient and of one of the two parents or holder of parental authority

Exclusion Criteria:

Inability to comply with the instructions defined and exposed during inclusion. Refusal of participation by the patient or one of the legal guardians

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * The patient presenting or having presented a TCA
  * The parents
  * One or more health professionals taking care of the patient
  * The school attended by the patient who will be questioned about the TCA and Covid-19 problem in general or not about the patient in particular.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Self-questionnaire Eating Attitudes Test-40 | at inclusion
  It is a self-diagnostic and quantitative questionnaire of 40 questions evaluating the behavior, severity and evolution of anorexia nervosa. The total score varies from 0 to 120. The threshold score is 30 to define an eating disorder

SECONDARY OUTCOMES:
Situational Anxiety and Trait Anxiety Inventory (STAI-Y) | at inclusion
  This inventory aims to assess anxiety as a "personality trait" (feelings of apprehension, tension, nervousness and worry that the subject usually feels), and anxiety as a ' "emotional state" linked to a particular situation (feelings of apprehension, tension or nervousness that the subject feels at a specific moment).
  This is a questionnaire comprising 20 items for the "state" form and 20 items for the "trait" form. The instruction is to answer "in general, in the usual way" for the "trait" scale and "at the moment" for the "state" scale.
  Each score can therefore vary from 20 to 80 with a "very high" anxiety norm when the threshold is > 65, "high" between 56 and 65, "medium" between 46 and 55, "low" between 36 and 45 and "very low" for a score < or = 35.
Beck Depression Inventory (BDI) scale | at inclusion
  The Beck Depression Inventory is a diagnostic self-questionnaire allowing a quantitative estimation of the intensity of depressive symptoms in adults and adolescents. It consists of 21 symptom and attitude items, which describe a specific behavioral manifestation of depression, graded from zero to three by a series of four statements reflecting the degree of severity of the symptom. The subject must indicate, among the propositions, the one that best describes how he has felt during the last seven days. The total score varies between 0 (absence of depressive symptoms) and 63. Some authors suggest that in a normal population, a total BDI score greater than 15 is an argument in favor of depression. The results of this scale can also be categorized according to: normal score < 15; mild depression: 10 to 18; moderate depression: 19 to 29; severe depression > 30.
Post-traumatic Check List Scale (PCL-5) | at inclusion
  The questionnaire includes 20 items, each question is to be rated between 1 and 5 depending on the intensity and frequency of symptoms during the previous month. The maximum score is 80. A threshold of 33 to 38 is proposed for screening for post-traumatic stress disorder (PTSD).

CONTACTS AND LOCATIONS:
Overall Officials: Louise-Emilie DUMAS, MD, Principal Investigator — Fondation Lenval
Locations (1):
- Hôpital Lenval, Nice, France